CLINICAL TRIAL: NCT04046653
Title: A Pre-biopsy Window of Opportunity Trial to Measure the Dietary Bioactive Levels in the Prostate Following an Intervention With Sulforaphane and Allin Dietary Supplements
Brief Title: Accumulation of Dietary Bioactives and Prostate Cancer
Acronym: ADaPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quadram Institute Bioscience (Other)
Collaborators: Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: QIB01/2019
Record Dates: First submitted 2019-07-17; First posted 2019-08-06 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — sulforaphane

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Study arm 1 (Experimental): Allin capsules (x2) and Sulforaphane capsules (x2) once daily for 4 weeks
  Interventions: Dietary Supplement: Allin; Dietary Supplement: Sulforaphane
- Study arm 2 (Experimental): Allin capsules (x2) and placebo capsules (x2) once daily for 4 weeks
  Interventions: Dietary Supplement: Allin; Dietary Supplement: Placebo
- Study arm 3 (Experimental): Sulforaphane capsules (x2) and placebo capsules (x2) once daily for 4 weeks
  Interventions: Dietary Supplement: Sulforaphane; Dietary Supplement: Placebo
- Study arm 4 (Placebo Comparator): Placebo capsules (x4) once daily for 4 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Allin — Dietary supplement
  Arms: Study arm 1; Study arm 2
Dietary Supplement: Sulforaphane — Dietary supplement
  Arms: Study arm 1; Study arm 3
Dietary Supplement: Placebo — Dietary supplement
  Arms: Study arm 2; Study arm 3; Study arm 4

SUMMARY:
Current research suggests that diets rich in multiple food types (such as broccoli, onions and garlic) are beneficial to our health and may reduce the risk of some cancers, including prostate cancer. The purpose of this study is to investigate the relationship between ingestion of the bioactive compounds from broccoli and garlic, and prostate metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for template biopsy of the prostate as part of routine investigation or staging for prostate cancer at the Norfolk and Norwich University Hospital
* BMI between 19.5 and 35 kg/m2
* Smokers and non-smokers

Exclusion Criteria:

* Those regularly taking 5α-reductase inhibitors or testosterone replacement medicines
* Those on warfarin treatment
* Those diagnosed with diabetes
* Those diagnosed with or suspected to be high-risk for human immunodeficiency virus (HIV) and/or viral hepatitis
* Those allergic to any of the ingredients included in the supplements (including those with lactose intolerance)
* Those taking additional dietary supplements or herbal remedies that could affect the study outcome.
* Those that are unable to understand English or give informed consent
* Parallel participation in another research project that involves dietary intervention
* Any person related to or living with any member of the study team.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2020-01-12 (Actual); Study Completion 2020-01-12 (Actual)

PRIMARY OUTCOMES:
Concentration of sulforaphane, alliin and their metabolites in prostate tissue as measured by mass spectrometry | 4 Weeks
  Treatment-related differences in prostatic accumulation of Sulforaphane and Alliin, or their human and microbial metabolites, compared with placebo following a 4-week period of supplementation

SECONDARY OUTCOMES:
2. Concentration of sulforaphane, alliin and their metabolites in in the transitional and peripheral zones of the prostate as measured by mass spectrometry | 4 weeks
  Treatment-related differences in spatial accumulation of Sulforaphane and Alliin, or their human and microbial metabolites, in the transitional and peripheral zones of the prostate compared with placebo following a 4-week period of supplementation
Urinary excretion of Sulforaphane and Alliin metabolites | 24-hours
  Treatment-related differences in the urinary excretion levels of Sulforaphane and Alliin, or their human and microbial metabolites, following the initial 24-h period of supplementation
4. Changes in global gene expression in prostate tissue as measured using next generation sequencing | 4 weeks
  Treatment-related differences in global gene expression in the prostate tissue, following a 4-week period of supplementation with Sulforaphane and Alliin, compared with placebo
Microbiome profile | 4 weeks
  Treatment-related differences in prostatic tissue microbiome from the peripheral and transitional zones, following a 4-week period of supplementation with Sulforaphane and Alliin compared with placebo
Number of participants with glutathione S-transferase M1 (GSTM1) genotype null and positive | After 4 weeks
  Changes in sulforaphane and alliin metabolites associated with Glutathione S-transferase M1 polymorphism (GSTM1 genotype)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Mithen, pHD, Principal Investigator — Quadram Institute Bioscience; Robert Mills, Dr, Principal Investigator — Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK)
Locations (1):
- Quadram Institute Bioscience, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: No